CLINICAL TRIAL: NCT00787475
Title: Northern Manhattan Diabetes Community Outreach Project
Acronym: NOCHOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Walter Palmas, MD, MS, FAHA, Associate Professor of Clinical Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAD1689; MD00206P60 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes
Keywords: Diabetes; Community health worker; Community outreach
MeSH Terms: conditions — Diabetes Mellitus | interventions — Community Health Workers

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): CHW intervention
  Interventions: Other: Community Health worker
- 2 (No Intervention): Enhanced usual care (brochure mailings)

INTERVENTIONS:
Other: Community Health worker — Community Health workers with at least 4 home visits, 8 phone calls, and 10 group visits.
  Arms: 1

SUMMARY:
The objective of this study is to examine the effectiveness of a community health worker intervention at helping to control diabetes among Latinos with poorly controlled Type 2 diabetes.

Hypothesis: Compared to those in Enhanced usual care group, patients randomized to the intervention will, at 12 months, have greater reductions in: (1) HgA1C; (2) low density lipoprotein (LDL); and (3) systolic and diastolic BP.

DETAILED DESCRIPTION:
The objective of this project is to examine the effectiveness of a community health worker (CHW) intervention at addressing glycemic control among Latinos with poorly controlled Type 2 diabetes. Our group has worked with a promising model of intervention that utilizes CHW's based at one of our major community partners. Pilot data from this program has shown clinically significant prepost test improvements in HgA1C. Using the Chronic Care Model as an overarching framework, the study design of NOCHOP is a randomized controlled trial of 360 Latinos, mostly of Caribbean descent, aged 35-70 years with HgA1C >=8.0. At a minimum, subjects in the intervention group will receive four home visits, ten group level visits and monthly phone calls by CHWs based at Alianza. The control groups will receive three separate mailings of bilingual diabetes health education materials. The primary outcome is glycemic control at 12month follow up, as measured by HgA1c. The secondary outcomes are changes in cholesterol and blood pressure (BP). We will also collect exploratory data on potential mechanisms through which our intervention resulted in hypothesized improvements including medication adherence, medication Intensification, diet and exercise. If successful, our project will make an important contribution to ongoing national and local debates about the sustainability of CHW programs. In particular, data from this study would be extremely useful for local Medicaid managed care plans who have expressed strong interests in data from rigorously designed clinical trials addressing the role of CHWs in delivering culturally appropriate and effective diabetes care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age 35-70 years*
* Receiving care at our clinic (2 visits with a primary care provider in the previous year)
* Living in Northern Manhattan or Western Bronx (based on zip codes)
* Had a hemoglobin A1C-done within the past year, with the latest value being > or = 8.0

Exclusion Criteria:

* Patients whose primary care physician (PCP) believes are not appropriate candidates for participation
* Type 1 diabetics (identified by PCP), as their care is quite distinct from that of Type II patients, and there are very few such patients in our clinic
* Patients with diabetes diagnosed when under age 25 ("new-onset" Type I diabetes) as such patients are extremely rare in our primary care clinics
* Patients who do not self-identify as Hispanic (Hispanics can be of any race e.g. white, black, mixed)
* Any life-threatening or extreme medical co-morbidity, such as an active cancer diagnosis, paraplegia, or end stage cardio-pulmonary disease
* Having a diabetes diagnosis for < 1 year, to ensure the stability of hemoglobin A1C values above 8.0
* Planning to move out of the neighborhood during the next year
* Planning to travel out of the neighborhood for more than three consecutive months
* Enrollment in any other cardiovascular disease (CVD) or diabetes intervention study

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2008-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
HgA1C level | Up to 12 months

SECONDARY OUTCOMES:
Measurement of LDL | Up to 12 months
Measurement of systolic blood pressure | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Walter Palmas, MD, Principal Investigator — Columbia University Medical Director
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Result] Palmas W, Findley SE, Mejia M, Batista M, Teresi J, Kong J, Silver S, Fleck EM, Luchsinger JA, Carrasquillo O. Results of the northern Manhattan diabetes community outreach project: a randomized trial studying a community health worker intervention to improve diabetes care in Hispanic adults. Diabetes Care. 2014 Apr;37(4):963-9. doi: 10.2337/dc13-2142. Epub 2014 Feb 4. PMID 24496805
- [Derived] Palmas W, Teresi JA, Findley S, Mejia M, Batista M, Kong J, Silver S, Luchsinger JA, Carrasquillo O. Protocol for the Northern Manhattan Diabetes Community Outreach Project. A randomised trial of a community health worker intervention to improve diabetes care in Hispanic adults. BMJ Open. 2012 Mar 26;2(2):e001051. doi: 10.1136/bmjopen-2012-001051. Print 2012. PMID 22454189